CLINICAL TRIAL: NCT02199015
Title: Lateral Cord Electrical Stimulation Can Improve Spasticity in Chronic Spastic Cerebral Palsy
Brief Title: Lateral Cord Stimulation as a New Treatment for Refractory Spastic Cerebral Palsy
Acronym: Andreani1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Carlos M. Andreani MD (Other)
Collaborators: Fundación CENIT (Unknown)
Responsible Party: Sponsor-Investigator, Juan Carlos M. Andreani MD, MD, Sociedad Argenttina de Neuromodulación
Organization: Sociedad Argenttina de Neuromodulación (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Andreani, JCM 1
Record Dates: First submitted 2014-07-17; First posted 2014-07-24 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy; Spasticity
Keywords: Dysarthria; Electrical Stimulation; Lateral Cord Stimulation; Spasticity; Treatment
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Spasticity, Cerebral Palsy (Experimental): To perform a Lateral spinal cord surgical implant of electrodes for electrical neuromodulation of a cohort of selectyed patients with refractory Spastic Cerebral Palsy To compare spasticity and speech trouble´s evolution on a cohort of treated patients, by evaluating their pre and post operative status into one year follow up.
  Interventions: Device: Lateral spinal cord surgical implant of electrodes

INTERVENTIONS:
Device: Lateral spinal cord surgical implant of electrodes — The procedure is based on the classic approaches to posterior cervical region for herniated discs, actually not longer employed for that aim A unilateral hemilaminectomy will be performed at C3-C4 level, starting from 4th cervical spinous process.
  A multicontact electrode will be placed on the lateral surface of the spinal cord that will be subcutaneusly connected to an implanted pulse generator (IPG).
  Other Names: Implant of Neurostimulators (electrical generators)

SUMMARY:
The aim of our work is to investigate whether electrical Lateral Cord Stimulation (LCS) causes an inhibitory and modulatory action by indirect cerebellar activation, so releasing spasticity and the spastic syndrome in selected cases of patients with cerebral palsy

DETAILED DESCRIPTION:
PROJECT Lateral Cord Stimulation was thought by the author to be employed in patients with spastic cerebral palsy with the aim to improve tonus, motor function and speech.

Nevertheless, as it has been demonstrated as acting on the basic phenomena related with spasticity, it's to say the propagated spinal responses, its use could be extended to other forms of spastic disease, like spastic limbs post stroke, brain congenital malformations producing spasticity and motor disorders as the main signs, post anoxic encephalopathy, etc.

In this preliminary clinical trial, classed as phase 3, our sample must be very limited to assure stable conditions for statistical significance, hence our group is going to be circumscribed to certain conditions and pathology.

In the future, as long the method could spread its use, the extension on indications in other pathological conditions is advisable thus, its possibilities of marketing could be enlarged with its use in a broader spectrum of spastic patients.

Calculated risks are similar to those related with the ancient surgical technique called "Scoville"technique, currently employed time ago for cervical discectomy (6) Investigational plan The purpose of this clinical trial is to release spasticity and by this means improve the condition of patients with spastic cerebral palsy by extradural lateral cord electrical stimulation, by using currently employed electrodes and neurostimulators Those devices are already FDA approved and currently used for Dorsal Column Stimulation with the objective to treat chronic Pain and spasticity (Spasmodic Torticollis).

ELIGIBILITY:
Inclusion Criteria:

* Aged sixteen or older
* Spastic Cerebral Palsy with stable condition
* Motor disability unilateral or predominantly unilateral.
* Troubles of speech clinically evident.
* Normal or Slightly sub-normal I.Q
* No psychiatric disorders.

Exclusion Criteria:

* Severe cardiac or respiratory troubles
* Fixed abnormal postures (except if previously corrected by orthopedic surgery)
* Chronic recurrent bronchial or pulmonary infections
* Chronic recurrent urinary infections
* Severe osteoporosis on affected limbs
* Chronic skin ulcerations.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Ashworth Scale | Day 0 baseline evaluation. One post operative evaluation every 30 day during six months
  The Ashworth scale has 5 points, they are: 1) no increase in muscle tone; 2) slight increase giving a catch when part is moved in flexion or extension; 3) more marked increase in tone but only after part is easily flexed; 4) considerable increase in tone; and 5) passive movement is difficult and affected part is rigid in flexion or extension

SECONDARY OUTCOMES:
Barthel Index | Day 0 baseline evaluation. One post operative evaluation every 30 day during six months
  The Barthel Index consists of 10 items that measure a person's daily functioning specifically the activities of daily living and mobility of the patient. The items include feeding, moving from wheelchair,etc, and the whole evaluation is from 100 maximum what means total independence, to 0, absolute dependence

OTHER OUTCOMES:
Functional Independence Measure (FIM)- for speech | Day 0 baseline evaluation. One post operative evaluation every 30 day during six months
  It is global independence assessment. In this case, we are going to take only those related to speech for disartria´s evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Andreani, MD, Study Director — Sociedad Argentina de Neuromodulación; Werner Braunsdorf, MD, Principal Investigator — Klinik von Magdeburg - Germany
Locations (2):
- Provincial Program of Neuromodulation, La Plata, Buenos Aires, Argentina
- Klinikummagdeburg, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Yes, we plan to share data as long as participants are recruited. Because there are not yet patients, we do not have data to share

REFERENCES:
- [Background] Andreani JC, Guma C. New animal model to mimic spastic cerebral palsy: the brain-damaged pig preparation. Neuromodulation. 2008 Jul;11(3):196-201. doi: 10.1111/j.1525-1403.2008.00166.x. PMID 22151096
- [Background] Andreani JC, Guma C. Lateral cord stimulation decreases spastic electromyographic spreading: responses in a brain-damaged pig preparation. Neuromodulation. 2008 Jul;11(3):202-7. doi: 10.1111/j.1525-1403.2008.00167.x. PMID 22151097